CLINICAL TRIAL: NCT01034163
Title: A Phase III Randomized, Double Blind, Placebo Controlled Multi-center Study of Panobinostat for Maintenance of Response in Patients With Hodgkin's Lymphoma Who Are at Risk for Relapse After High Dose Chemotherapy and Autologous Stem Cell Transplant (ASCT)
Brief Title: A Phase III Randomized, Double Blind, Placebo Controlled Multi-center Study of Panobinostat for Maintenance of Response in Patients With Hodgkin's Lymphoma (HL)
Acronym: PATH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBH589E2301; 2009-014846-26
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-05

CONDITIONS: Hodgkin's Lymphoma
Keywords: Phase III randomized; double blind; placebo controlled multi-center study; panobinostat; Hodgkin's lymphoma; at risk for relapse; autologous stem cell transplant
MeSH Terms: conditions — Hodgkin Disease | interventions — Panobinostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panobinostat (PAN) (Experimental): Participants received 45 mg orally 3 times a week (TIW), every other week (QOW),
  Interventions: Drug: Panobinostat
- Placebo (Placebo Comparator): Participants received matching placebo to PAN TIW, QOW.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Panobinostat
  Other Names: LBH589
  Arms: Panobinostat (PAN)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective was to provide drug to ongoing patients who were receiving panobinostat and to characterize the safety and tolerability of panobinostat in patients with HL after achieving a complete response following autologous hematopoietic stem cell transplant (AHSCT) with high dose chemotherapy (HDT). Primary objective as stated above reflects a change from the original protocol as of an amendment. The original objective was no longer feasible with only 41 of 367 patients randomized after the study was halted due to poor recruitment. An amendment was written to allow patients on panobinostat to continue their treatment until discontinuation/completion criteria were met (patients were unblinded). Therefore, the study was completed as per this amendment. No secondary objectives were included for this trial from the amendment; this was a change from the original protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is greater than or equal to 18 years
2. Patient has a history of histologically confirmed classical HL (i.e. Nodular sclerosing (NSHL), Mixed-cellularity (MCHL), Lymphocyte-rich (LRHL), Lymphocyte depleted (LDHL))
3. Patient has achieved a complete response by CT/MRI scan within 9 weeks (± 1 week) from the day of their first autologous peripheral blood/ bone marrow stem cell transfusion (AHSCT) following HDT. Complete response is defined as:

   Normalization of all nodes and lesions compared to pre-transplant scan performed prior to salvage therapy for relapse. Any residual abnormal masses on the post transplant CT/MRI must be metabolically inactive on a PET scan.
4. Patient has at least one of the following factors that places them at risk for relapse:

   * Primary refractory disease (including relapse in ≤ 3 months of completion of 1st line treatment)
   * First relapse >3 but <12 months from last dose of 1st line treatment
   * Multiple relapses (prior to transplant)
   * Stage III/IV disease (at relapse, prior to transplant)
   * Hemoglobin <10.5 gm/dL (at relapse, prior to transplant)

Exclusion Criteria:

Patient has been treated with allogeneic transplant 2. Patient has received any anti-lymphoma therapy after AHSCT including but not limited to:

* chemotherapy prior to start of study
* biologic immunotherapy including monoclonal antibodies or experimental therapy prior to start of study
* radiation therapy 3. Patient has not recovered from reversible toxicity due to any prior therapies (e.g. returned to baseline or Grade ≤1) except for hematological laboratory parameters Note: Patient does not meet this criteria if the toxicity is stable and irreversible, and there is no evidence that panobinostat causes a similar toxicity 4. Patient has received prior treatment with DAC inhibitors including panobinostat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- United States (13):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - Georgia Health Sciences University Medical College of Georgia, Augusta, Georgia
  - Northwestern University Oncology, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester Hematology/Oncology Dept., Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina Oncology, Charleston, South Carolina
  - Vanderbilt University Medical Center Vanderbilt Clinic - Oncology, Nashville, Tennessee
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Medical College of Wisconsin Oncology, Milwaukee, Wisconsin
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Brazil (2):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (3):
  - Novartis Investigative Site, Caen, Cedex
  - Novartis Investigative Site, Lille, France
  - Novartis Investigative Site, Dijon
- Germany (3):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Essen-Werden
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
- Novartis Investigative Site, Reggio Calabria, RC, Italy
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Christchurch, New Zealand
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Wroclaw
- Russia (2):
  - Novartis Investigative Site, ChelyabinskChemo
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 2:1 ratio to the PAN and placebo groups, respectively.
Groups:
- Panobinostat (PAN): Participants received 45 mg orally 3 times a week (TIW), every other week (QOW).
Period: Overall Study
Arm/Group | Panobinostat (PAN) | Placebo
Started | 27 | 14
Untreated (Not in Safety Set) | 1 | 2
Safety Set | 26 | 12
In Open Label Phase After Unblinding | 5 | 0
Completed | 0 | 0
Not Completed | 27 | 14
Not completed — Treatment completed as per protocol | 8 | 7
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Protocol deviation | 1 | 0
Not completed — Disease progression | 3 | 4
Not completed — Adverse Event | 6 | 0
Not completed — Administrative problems | 0 | 1
Not completed — Abnormal laboratory value | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panobinostat (PAN) | Placebo | Total
Number analyzed (Participants) | 27 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (10.72) | 30.6 (10.56) | 32.9 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 19 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Safety monitoring was conducted throughout the study.
Time Frame: 23 months
Population: Safety set: The safety set included randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Panobinostat (PAN) | Placebo
Number analyzed (Participants) | 26 | 12
Participants | 26 | 11

ADVERSE EVENTS:
Arm/Group | Panobinostat (PAN) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/12
Other Adverse Events (participants affected / at risk) | 26/26 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (PAN) (N=26) | Placebo (N=12)
Pyrexia (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Sinusitis bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (PAN) (N=26) | Placebo (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 7 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 23 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 15 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 12 | 3
Asthenia (General disorders) | 3 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 9 | 3
Influenza like illness (General disorders) | 4 | 0
Mucosal dryness (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 1
Swelling (General disorders) | 0 | 1
Herpes ophthalmic (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 0
Oral infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Blood triglycerides increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 6 | 0
Polyneuropathy (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.